CLINICAL TRIAL: NCT06914739
Title: Application of Health Empowerment Theory to Enhance Health Empowerment Levels and Self-Health Management Ability Among Older Migrants: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TianLe Xiang (Other)
Responsible Party: Sponsor-Investigator, TianLe Xiang, postgraduate, Huzhou University
Organization: Huzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2022011
Record Dates: First submitted 2025-03-31; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Health Self-management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An researcher uninvolved in the enrollment or the intervention organized the randomization. The HET-based program providers who performed the intervention were not blinded, as the intervention was based on HET-based program, which is different from regular care. However，those assessing the intervention outcome were blinded from group assignment for the majority of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The intervention group (Experimental): The intervention group received the HET-based intervention program for 12 weeks.
  Interventions: Behavioral: The Health Empowerment Theory (HET) program
- routine community care (Active Comparator): The control group received routine community care for 12 weeks.
  Interventions: Behavioral: routine community care

INTERVENTIONS:
Behavioral: The Health Empowerment Theory (HET) program — The intervention group received the HET-based intervention program for 12 weeks. From the first week to the fourth week, community nurses interacted with the participants face-to-face to analyze and establish their problems and needs in health management (usual community health services utilization, such as medicine purchases and vaccinations) and helped clarify the importance of health management and their strengths (such as existing health knowledge). From the fifth to twelfth weeks, participants attended health knowledge lectures led by community nurses, covering topics such as: a) healthy lifestyle, primarily diet, exercise, and disease prevention and management for older adults; and b) community health services, which included recent or long-term community health services (such as health examinations for older adults and family doctor contracts). WeChat groups and offline gatherings at community health centers (with groups of eight to ten peers) were organized to interact and comm
  Arms: The intervention group
Behavioral: routine community care — The control group received routine community care, including notifications of community- related activities and lectures through WeChat group chats or telephone calls, and had questions answered by researchers and community nurses.
  Arms: routine community care

SUMMARY:
This study aimed to evaluate the effectiveness of a theory-based health self-management program in empowering older migrants to manage their health. This study used a single-blind, randomized controlled trial design. A comparison was conducted between the experimental and control groups in terms of pre-test and post-test levels of health empowerment and health self-management abilities.

ELIGIBILITY:
Inclusion Criteria:

* (1) age 60 years or older; (2) residing in thelocal area for a minimum of six months; (3) agreement to participate in the study and willingness tosign the informed consent form; and (4) possessing a clear sense of autonomy and the ability tounderstand and engage with the content of the study intervention activities.

Exclusion Criteria:

* (1) absencefrom two consecutive lectures or group activities without prior notification and (2) voluntary withdrawal from the study at the participant's request.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
health empowerment level | From enrollment to the end of treatment at 12 weeks
  The Older Health Empowerment Evaluation Scale comprises six subdimensions: liability beliefs, knowledge and skills, external support, participation in health management, acceptance of change, and empowerment of others.35 The scale consists of 38 items. A Likert 5-point scoring method was employed, with a total score ranging from 38 to 190. A high score indicates a high level of health empowerment among older adults. The total Cronbach's α coefficient was 0.959, with the Cronbach's α coefficient of each dimension ranging from 0.827 to 0.890. This scale was used to replace the chronic disease older health empowerment scale, mainly to better assess health empowerment in older adults and reflect subtle but significant differences in empowerment levels between the older groups.

SECONDARY OUTCOMES:
self-health management ability | From enrollment to the end of treatment at 12 weeks
  The Adult Health Self-Management Skill Rating Scale is a widely used instrument for evaluating individual self-health management ability.36 The formal scale consists of three subscales with 38 items: the Health Self-Management Cognition subscale (14 items), Self-Management Environment subscale (10 items), and Health Self-Management Behavior subscale (14 items). A Likert 5-point scoring method was employed, whereby a high score indicates a high level of health self-management ability. A score of 36 to 76 indicates a low level of ability, 77 to 152 denotes a medium level, and 153 to 190 indicates a high level of ability. The Cronbach's α coefficient of the scale was 0.993, and the content validity was 0.895.

CONTACTS AND LOCATIONS:
Locations (1):
- Huzhou University, Huzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No